CLINICAL TRIAL: NCT00597649
Title: An Open-Label 52-Week Safety Study of Bicifadine SR in Adult Outpatients With Chronic Peripheral Neuropathic Pain Associated With Diabetic Peripheral Neuropathy
Brief Title: A 52-Week Study of Bicifadine in Patients With Chronic Neuropathic Pain Associated With Diabetic Peripheral Neuropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The 001 trial did not show benefit versus placebo
Sponsor: XTL Biopharmaceuticals (Industry)
Responsible Party: Mark Roffman, Vice President, XTL Biopharmaceutical Co.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XTL B07-002; 2007-003638-40
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Chronic Peripheral Neuropathy Pain in Diabetics
MeSH Terms: interventions — bicifadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Bicifadine 800 mg/day for a year
  Interventions: Drug: Bicifadine
- 2 (Experimental): Bicifadine 1200 mg/day for a year
  Interventions: Drug: Bicifadine

INTERVENTIONS:
Drug: Bicifadine — SR dosage form of 400 mg bid or tid for one year

SUMMARY:
This study is to evaluate the long-term efficacy and safety of two dosages of bicifadine SR (600 mg/day and 1200 mg/day) for up to 52 weeks in reducing chronic peripheral neuropathy pain due to diabetes in adult outpatients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years or older
* Diagnosis of type 1 or type 2 non-insulin dependent diabetes mellitus
* Chronic bilateral pain due to diabetic neuropathy, pain for at least six months.
* Primary pain is located in the feet.
* Subject participated in and completed the XTL 07-001 clinical trial.

Contact site for additional information.

Exclusion Criteria:

* Symptoms of other painful conditions
* Presence of amputations other than toes
* Clinically significant psychiatric or other neuropsychological disorder
* Use of certain medications
* Clinically important other diseases
* Pregnancy
* History of alcohol or narcotic abuse within two years.

Contact site for additional information.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pain and safety | one year

SECONDARY OUTCOMES:
Clinical Global Impression of Improvement; McGill Pain Questionnaire; Amount of Rescue Medication Used for Pain; Quality of Life Survey (SF-36); Patient Global Impression of Change | One year

CONTACTS AND LOCATIONS:
Overall Officials: Mark Roffman, PhD, Study Director — XTL Biopharmaceuticals
Locations (1):
- Four Rivers Clinical Research, Paducah, Kentucky, United States

REFERENCES:
- See also: Sponsor's website — http://www.xtlbio.com